CLINICAL TRIAL: NCT04546763
Title: Study Watch AF Detection At Home
Status: Completed | Type: Observational
Sponsor: Verily Life Sciences LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 102238
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Paroxysmal Atrial Fibrillation Patients: This will be a single arm study of patients with paroxysmal atrial fibrillation. Subjects will be wearing the Study Watch and Zio XT Patch concurrently for up to 14 days.
  Interventions: Device: Study Watch; Device: Zio XT

INTERVENTIONS:
Device: Study Watch — The Study Watch is a miniaturized wearable device made with biocompatible contact materials containing various sensors capable of measuring physiological and environmental metrics.
Device: Zio XT — The Zio XT Patch, the reference device, is a FDA-cleared single-patient use, continuously recording ECG monitor that can be worn up to 14 days.

SUMMARY:
This is a multi-center, prospective, non-randomized study to evaluate the performance of the study watch PPG algorithm in detecting irregular rhythms suggestive of atrial fibrillation (AF) in subjects at risk of having an event of AF in the free living (home) environment.

ELIGIBILITY:
Inclusion Criteria:

* At least 22 years old
* Able to read and speak English
* Able and willing to sign written Informed Consent
* Interest in participating in the study
* At risk of having an AF event, as determined by having a diagnosis of paroxysmal AF (PAF) and meeting one of the following: (a) scheduled or to be scheduled to undergo AF ablation, (b) with implantable loop recorder (ILR), implantable cardioverter defibrillator (ICD), permanent pacemaker (PPM), holter monitor, or adhesive monitoring patch with documented AF burden of ≥25% in the 3 months prior to consent date, (c) CHA2DS2VASc ≥3, (d) Left atrial diameter ≥4.4 cm
* Without significant limitation in ability to participate in the study, in the opinion of the investigator

Exclusion Criteria:

* Currently in a paced rhythm
* Currently on class Ic or class III antiarrhythmic medication that has been successful in eliminating AF (no documented AF of more than 30 seconds since the initiation of the medication)
* Had successful AF ablation (no documented AF of more than 30 seconds post procedure)
* Known severe allergy to nickel or metal jewelry
* Known allergic reaction to adhesives or hydrogels or with family history of adhesive skin allergies
* Are diagnosed with persistent AF
* Use of implantable neuro-stimulator
* Open injury or rash where the study device or comparator will be worn

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At risk of having an AF event, as determined by having a diagnosis of paroxysmal AF (PAF)
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Accuracy of AF detection - Sensitivity | 14 days
  Accuracy of AF detection based on sensitivity observed in a 14-day followup period
Accuracy of AF detection - Specificity | 14 days
  Accuracy of AF detection based on specificity observed in a 14-day followup period

SECONDARY OUTCOMES:
A sensitivity analysis estimating the range of sensitivities | 14 days
  A sensitivity analysis estimating the range of sensitivities when imputing insufficient quality data
A sensitivity analysis estimating the range of specificities | 14 days
  A sensitivity analysis estimating the range of specificities when imputing insufficient quality data
Estimates of sensitivity by protocol-defined subgroups | 14 days
  Estimates of sensitivity by protocol-defined subgroups
Estimates of specificity in subgroups | 14 days
  Estimates of specificity in subgroups defined by: race, age-groups, site, activity levels, and AF-burden
Estimates of positive predictive value (PPV) on the AF-burden | 14 days
  Estimates of PPV based on the AF-burden observed in the study
Estimates of negative predictive value (NPV) on the AF-burden | 14 days
  Estimates of NPV based on the AF-burden observed in the study
Estimates of PPV on the AF burden to a screening population | 14 days
  Estimates of PPV based on the AF burden relevant to a screening population
Estimates of NPV on the AF burden to a screening population | 14 days
  Estimates of NPV based on the AF burden relevant to a screening population

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Ghanbari, Principal Investigator — Verily Life Sciences
Locations (5):
- United States (5):
  - San Diego Cardiac Center, San Diego, California
  - Colorado Heart and Vascular, Lakewood, Colorado
  - Ascension Providence Hospital, Southfield, Michigan
  - UPMC Pinnacle Harrisburg, Harrisburg, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Poh MZ, Battisti AJ, Cheng LF, Lin J, Patwardhan A, Venkataraman GS, Athill CA, Patel NS, Patel CP, Machado CE, Ellis JT, Crosson LA, Tamura Y, Plowman RS, Turakhia MP, Ghanbari H. Validation of a Deep Learning Algorithm for Continuous, Real-Time Detection of Atrial Fibrillation Using a Wrist-Worn Device in an Ambulatory Environment. J Am Heart Assoc. 2023 Oct 3;12(19):e030543. doi: 10.1161/JAHA.123.030543. Epub 2023 Sep 26. PMID 37750558